CLINICAL TRIAL: NCT00411996
Title: The Pharmacokinetics and Safety of Ritonavir-boosted Indinavir 600/100mg Bid Combined With NRTIs in ARV naïve HIV/TB Co-infected Patients Receiving Rifampicin Containing Anti-tuberculosis Therapy
Brief Title: The Pharmacokinetics and Safety of IDV/r With NRTIs in HIV/TB Co-infected Patients Receiving Rifampicin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 044
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: indinavir/ritonavir; HIV/TB; rifampicin; PK and efficacy of IDV/RTV 600/100 mg BID with rifampicin; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Indinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): IDV/r 600/100 mg + rifampicin
  Interventions: Drug: indinavir/ritonavir

INTERVENTIONS:
Drug: indinavir/ritonavir — IDV/r 600/100 mg BID + rifampicin OD for at least 2 weeks

SUMMARY:
We believe that there is a strong rationale for the study of IDV/r 600/100 bid as a boosted-PI combination that, in the presence of RMP, is able to produce a satisfactory PK profile associated with adequate antiretroviral potency, tolerability and efficacy.

DETAILED DESCRIPTION:
The fixed-dose combination of d4T+3TC+NVP (GPOvir) has been widely used in Thailand since June 2002. The prevalence of NNRTI resistance has increased since 2005. Efavirenz-based antiretroviral therapy (ART) is preferred in patients with TB/HIV receiving rifampin-containing TB regimens. However, efavirenz cannot be used in the context of NNRTI failure, intolerance or toxicity. The optimal ART in populations receiving rifampicin remains unknown. Rifabutin, which is recommended in combination with a boosted protease inhibitor (PI/r) is expensive and not available in Thailand and other developing countries. Ritonavir-boosted indinavir (IDV/r) is potent and the cheapest boosted PI available in Thailand. If IDV/r in combination with rifampin demonstrates suitable pharmacokinetics and is well tolerated, this regimen might prove useful and could be widely implemented. However, high rates of gastrointestinal and renal toxicity have been demonstrated in Thai patients receiving standard doses of IDV/r 800/100 BID. We believe that there is a strong rationale to study if IDV/r 600/100 BID in combination with rifampin is able to produce a satisfactory pharmacokinetic profile, with antiretroviral potency, tolerability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV positive after voluntary counselling and testing
* Aged between 18 and 60 years of age
* Antiretroviral treatment naive
* CD4+ cell count of <200 cells/mm3 at the time of TB diagnosis
* ALT <5 times ULN
* Serum creatinine <1.4 mg/dl
* Haemoglobin >8 mg/L
* TB diagnosis; either probable (clinical symptoms plus chest x-ray and response to anti-TB medication) or definitive( sputum AFB culture confirmed) and receiving or planning to receive rifampicin-containing anti-TB therapy for at least a 2 week period before the initiation of ART
* No other active OI (CDC class C event)
* Able to provide written informed consent

Exclusion Criteria:

* Current use of steroids and other immunosuppressive agents
* Current use of any prohibited medications related to compliance and drug pharmacokinetics
* Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the trial.
* Previous exposure to nevirapine monotherapy
* Unlikely to be able to remain in follow-up for the protocol defined period
* Patients with proven or suspected acute hepatitis. Patients with chronic viral hepatitis are eligible provided ALT, AST < 5 x ULN.
* Karnofsky performance score <30%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of ritonavir-boosted indinavir 600/100mg bid in combination with rifampicin-containing anti-TB therapy. | 2 weeks

SECONDARY OUTCOMES:
safety of ritonavir-boosted indinavir 600/100mg bid in combination with rifampicin-containing anti-TB therapy | 48 weeks
efficacy of ritonavir-boosted indinavir 600/100mg bid in combination with rifampicin-containing anti-TB therapy | 48 weeks
the prevalence of immune recovery syndrome of TB and other HIV-related conditions after ritonavir-boosted indinavir 600/100mg bid | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT, Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- [Derived] Avihingsanon A, van der Lugt J, Singphore U, Gorowara M, Boyd M, Ananworanich J, Phanuphak P, Burger D, Ruxrungtham K. Pharmacokinetics and 48 week efficacy of adjusted dose indinavir/ritonavir in rifampicin-treated HIV/tuberculosis-coinfected patients: a pilot study. AIDS Res Hum Retroviruses. 2012 Oct;28(10):1170-6. doi: 10.1089/AID.2011.0247. Epub 2012 Mar 6. PMID 22250979
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org